CLINICAL TRIAL: NCT00507598
Title: Metabolomics-Based Detection of Colorectal Cancer
Acronym: metabolomics
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 0706-03: IUCRO-0198
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; metabolomics
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, urine
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — Correlative study collecting serum and tissue samples

SUMMARY:
The purpose of this study is to collect specimens to perform metabolic profiling of serum and urine from patients with colorectal cancer, colon polyps and healthy patients.

DETAILED DESCRIPTION:
In this study, metabolite profiling analysis will be carried out on colon cancer patients at the time of diagnosis and during the course of treatment, using patient tissue and serum samples. Samples of serum (1 ml) and tissue specimens (50 mg each) from colorectal cancer patients (stages I-IV) and serum samples from an equal number of age and gender-matched healthy controls will be obtained under identical (8-hour overnight fasting) conditions. Metabolic profiles will be identified using the NMR and MS instruments located in Purdue's on-campus NMR and MS facilities. Multivariate statistical analyses will be used to monitor changing metabolite profiles that indicate changes in disease status. We anticipate that putative biomarkers will be easier to identify in the cancerous tissue, and the concentrations of these metabolites will then be quantified in the patients' serum, that ultimately would allow for easier detection of colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resectable colorectal cancer must have samples collected (serum/urine) prior to surgery and/or after surgery, but prior to starting chemotherapy.
* Patients with metastatic colorectal cancer must have samples collected prior to initiating chemotherapy, and after chemotherapy initiation: every 3 months for up to 24 months.
* Subjects must be ≥ 18 years of age.
* Subjects undergoing screening colonoscopy are able to participate as healthy controls or as patients with colon polyps if colonoscopy identifies colon polyps being present (informed consent will be signed first and samples will be collected; after colonoscopy the samples will be identified as "healthy" or "polyps").
* For patients who underwent biopsy or surgery for colorectal cancer, enough tissue needs to be available for testing, as appropriate per patients groups in the protocol Schema.
* Subjects must be able to attend follow up or treatment visits per investigator's recommendations for up to 24 months for collection of serum/urine specimens.
* Female patients known to be pregnant are not eligible for this protocol.
* Subjects must be able to undergo an 8-hr overnight fast prior to metabolomic testing

Exclusion Criteria:

* Presence of an invasive cancer other than colorectal cancer is an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: colorectal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
•Perform metabolic profiling of tissue,serum & urine from pts w/ colorectal cancer (stages I-IV), healthy controls & pts w/ colorectal polyps & correlate results. | 1 years

SECONDARY OUTCOMES:
Correlate changes of serum & urine biomarkers /p trt to predict response or toxicity,& correlate w/other treatment outcomes. Compare the metabolic profile between pts w/various stages of colorectal cancer. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elena Chiorean, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States